CLINICAL TRIAL: NCT02290509
Title: Double-Blind, Randomized, Active-Controlled Comparison of the Immunogenicity and Safety of Flublok® Quadrivalent Versus IIV4 in Healthy, Medically Stable Adults 18-49 Years of Age
Brief Title: Safety and Immunogenicity of Flublok Quadrivalent vs IIV4 in Adults 18-49 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Collaborators: Syneos Health (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSC16
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flublok Quadrivalent Influenza Vaccine (Experimental): Intramuscular injection of vaccine containing 4 x 45µg (180µg total) of each recombinant hemagglutinin (rHA) derived from influenza A/H1N1 and A/H3N2 and two lineages of influenza B viruses identified for the season in which the trial is conducted in a total volume of 0.5 mL
  Interventions: Biological: Flublok Quadrivalent
- Inactivated Influenza Vaccine (IIV4) (Active Comparator): Intramuscular injection of vaccine contains 4 x 15µg (60µg total) of HA derived from the same influenza A/H1N1 and A/H3N2 and influenza B strains in a total volume of 0.5mL.
  Interventions: Biological: Inactivated Influenza Vaccine (IIV4)

INTERVENTIONS:
Biological: Flublok Quadrivalent — Intramuscular injection of study vaccine
  Arms: Flublok Quadrivalent Influenza Vaccine
Biological: Inactivated Influenza Vaccine (IIV4) — Intramuscular injection of study vaccine
  Arms: Inactivated Influenza Vaccine (IIV4)

SUMMARY:
Randomized, double-blind trial of safety and immunogenicity of Flublok Quadrivalent versus Inactivated Influenza Vaccine (IIV4) in 1350 healthy, medically stable adults 18-49 years of age. Serum samples for Hemagglutinin Inhibition titers will be determined pre- and 28 days post-vaccination. Subjects will be followed for 6 months after vaccination for serious and/or medically-attended adverse events.

DETAILED DESCRIPTION:
As the spectrum of influenza vaccines rapidly evolves to quadrivalent formulations with the intention of offering broader protection to include both lineages of influenza B strains, it is appropriate to transition Flublok from a trivalent to a quadrivalent formulation. The demonstration of non-inferior post-vaccination Hemagglutination Inhibition Assay (HAI) Geometric Mean Titers (GMTs) to antigens in the Flublok Quadrivalent formulation compared to those of the matching antigens in a US - approved IIV4 is intended to support licensure of Flublok Quadrivalent for the adult population for which Flublok trivalent is currently approved. The comparison of safety and reactogenicity of Flublok Quadrivalent to that of IIV4 is expected to confirm a similar safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, in good health or medically stable
* Able to understand and comply with planned study procedures
* Provide written informed consent
* Negative urine pregnancy test within 24 hours prior to vaccination (women of child-bearing potential)

Exclusion Criteria:

* Prior serious or severe reaction to influenza vaccine
* Known contraindication to either study vaccine
* Receipt of any other influenza vaccine within 180 days prior to enrollment
* Plan to receive another licensed influenza or other vaccine during the duration of this study
* Receipt of any significant new diagnosis, medication (licensed or investigational), or licensed vaccine within 30 days prior to enrollment in this study
* Underlying disease or therapeutic intervention that might adversely affect the immune response
* Plans to participate in any investigation involving an investigational product during this study.
* Pregnant, lactating or planning to become pregnant within 30 days of study vaccine.
* Any clinical or social circumstance that in the opinion of the investigator could interfere with compliance with study procedures or interfere with the interpretation

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1350 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Seger, MD, Principal Investigator — Benchmark Research, Fort Worth, TX
Locations (10):
- United States (10):
  - Benchmark Research - Sacramento, Sacramento, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Meridian Research, Bellevue, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Meridian Research, Dakota Dunes, South Dakota
  - Benchmark Reseach, Austin, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas

REFERENCES:
- [Derived] Dunkle LM, Izikson R, Patriarca PA, Goldenthal KL, Muse D, Cox MMJ. Randomized Comparison of Immunogenicity and Safety of Quadrivalent Recombinant Versus Inactivated Influenza Vaccine in Healthy Adults 18-49 Years of Age. J Infect Dis. 2017 Dec 5;216(10):1219-1226. doi: 10.1093/infdis/jix478. PMID 28968871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Started | 1011 | 339
Completed | 962 | 325
Not Completed | 49 | 14

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes the Safety Population, all randomized subjects who were immunized and provided any safety data (solicited or unsolicited) following administration of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4) | Total
Number analyzed (Participants) | 998 | 332 | 1330
Age, Customized [Number; unit: participants]
  18-49 years | 998 | 332 | 1330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 639 | 222 | 861
  Male | 359 | 110 | 469
Region of Enrollment [Number; unit: participants]
  United States | 998 | 332 | 1330

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion to Vaccine Antigens Following Vaccination With Quadrivalent Vaccine
Description: Seroconversion is defined as: Either a pre vaccination titer < 10 (1/dil) and a post vaccination titer ≥ 40 (1/dil), or a pre vaccination titer ≥ 10 (1/dil) and a ≥ 4 fold increase in post vaccination titer at Day 28 after the final vaccination.
Time Frame: Day 28 after final vaccination
Population: The immunogenicity population includes all randomized subjects who received a dose of study vaccine, provided serum samples for baseline (Day 0) and Day 28 HAI titers (within the specified windows) and have no major protocol deviations that might have adversely affect the immune response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 969 | 323
percentage of participants
  A/H1N1/California | 66.7 [63.6 to 69.6] | 63.5 [58.0 to 68.7]
  A/H3N2/Texas | 72.1 [69.2 to 74.9] | 57.0 [51.4 to 62.4]
  B/Massachusetts | 59.6 [56.5 to 62.8] | 60.4 [54.8 to 65.7]
  B/Brisbane | 40.6 [37.4 to 43.7] | 58.2 [52.6 to 63.6]

2. Secondary Outcome: Number of Participants With Systemic and Injection Site Reactogenicity
Time Frame: Days 0-7
Population: The Reactogenicity Population includes subjects who recorded any systemic reaction data and injection site reaction data following administration of study vaccine. This was two subjects less than the Safety Population.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 996 | 332
participants
  Subjects with one or more injection site reaction | 510 | 172
  Subjects with one or more systemic reaction event | 339 | 119

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Medically-attended Adverse Events (MAEs)
Time Frame: Six months post-vaccination
Population: The safety population includes all randomized and vaccinated subjects who provided any safety data (solicited or unsolicited) following administration of study vaccine.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 998 | 332
participants
  Serious adverse events (SAEs) | 10 | 2
  Medically-attended adverse events (MAEs) | 80 | 24

4. Primary Outcome: Geometric Mean Titers of Antibodies to Vaccine Antigens Following Vaccination With Quadrivalent Vaccine
Description: Immunogenicity will be evaluated prior to vaccination and at 28 days after vaccination using the hemagglutination inhibition (HAI) technique. For each influenza vaccine strain, pre and post vaccination geometric mean titers (GMTs) were calculated.
Time Frame: Day 0 and Day 28 after final vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Number analyzed (Participants) | 969 | 323
titer
  Day 0 - A/H1N1/California | 60 [54 to 65] | 54 [46 to 63]
  Day 28 - A/H1N1/California | 502 [469 to 537] | 407 [367 to 451]
  Day 0 - A/H3N2/Texas | 75 [68 to 83] | 70 [60 to 82]
  Day 28 - A/H3N2/Texas | 757 [709 to 808] | 385 [348 to 425]
  Day 0 - B/Massachusetts | 27 [25 to 29] | 24 [21 to 28]
  Day 28 - B/Massachusetts | 159 [147 to 171] | 136 [121 to 153]
  Day 0 - B/Brisbane | 12 [11 to 13] | 11 [10 to 12]
  Day 28 - B/Brisbane | 43 [40 to 46] | 64 [58 to 72]

ADVERSE EVENTS:
Time Frame: All AEs collected 28 days after study immunization and all Serious Adverse Events (SAEs) collected through six (6) months after study immunization.
Description: The safety population includes all randomized and vaccinated subjects who provided any safety data (solicited or unsolicited) following administration of study vaccine.
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine (IIV4)
Serious Adverse Events (participants affected / at risk) | 10/998 | 2/332
Other Adverse Events (participants affected / at risk) | 63/998 | 24/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok Quadrivalent Influenza Vaccine (N=998) | Inactivated Influenza Vaccine (IIV4) (N=332)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Periumbilical abcess (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Arm amputation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok Quadrivalent Influenza Vaccine (N=998) | Inactivated Influenza Vaccine (IIV4) (N=332)
Nasophayngitis (Infections and infestations) | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 10 | 5
Sinusitis (Infections and infestations) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Headache (Nervous system disorders) | 20 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less